CLINICAL TRIAL: NCT00521287
Title: Adjustment of Optimal Immune System by Using Cytokine Cocktails Before Applying DC Vaccine
Brief Title: Impaired Immunity in Patients With Cancer: Influence of Cancer Stage, Chemotherapy, and Cytomegalovirus Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Yen Ta Lu/ Dr., Mackay Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MMH-I-S-321; MMH-I-S-401
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2007-08

CONDITIONS: Neoplasms
Keywords: Immunologic Surveillance; Vaccination; Immunotherapy; Dendritic Cells
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early (E) (Other): Early stage cancer
  Interventions: Other: Immune profiling and DC vaccine
- Advanced (A) (Other): Advanced stage cancer (Stage IV without treatment)
  Interventions: Other: Immune profiling and DC vaccine
- Terminal (T) (Other): Terminal stage cancer (Stage IV with chemotherapy)
  Interventions: Other: Immune profiling and DC vaccine

INTERVENTIONS:
Other: Immune profiling and DC vaccine — 1. For observational study (immune profiling): blood sampling 3-5 mL
  2. For DC vaccine: one dose of DC vaccine(~10 million cells)/2 week for at least 6 month or until progression.
  Other Names: cytokine cocktail

SUMMARY:
According to a survey from Department of Health in 2004, cancer has been the leading cause of death in the Taiwan area. In 2004, people died of cancer, accounting for 27.2 percent of all deaths. The major reason of the superior grade is that cancer has the ability to escape the surveillance of immune system. It is also a main issue to address in medical research.

Dendritic cells (DCs), the most potent APC, are located at sites of pathogen entry, acquire antigens from pathogens or pathogen-infected cells, and process these antigens for both class I and class II presentation. Upon antigen encounter, they termed immature DCs, undergo a maturation process, they are capable to present captured antigens to T cells. This maturation step allows DC migration to trigger adaptive immune responses. These features make DCs very good candidates for therapy against various pathological conditions including malignancies.

Therefore, two concepts in this project will be concerned: one is enhancement of T cell immunity and the other is improvement of the efficiency of DC-tumor fusion. The strategy of enhance T cell is using well-known cytokines, such as IL2, and IL7 to expand the tumor-specific CD4 and CD8 T cells before DC-vaccine treatment. In the past, scientists utilized polyethyleneglycol to fuse cancer cells and dendritic cells. However, the results were devastating. Two new approaches of the DC vaccine will be applied to this study: DC-tumor fusion and DC phagocytosed apoptosed tumor cells. Whole tumor cells will be fused with DCs by combining hypotonic buffer and electrical-based fusion protocols. The safety of hybrid cell vaccination has been shown in clinical trials with some encouraging anti-tumour effects. However, data are as yet insufficient to assess a clear therapeutic benefit. Hopefully, the combination of two strategies will improve the efficiency of DC vaccine and boost survival of cancer patients.

As we have gained a clearer understanding of the cellular and molecular events that modulate antigen presentation and T cell activation in vivo, new strategies have emerged, allowing the development of more potent second generation DC vaccines.

ELIGIBILITY:
Inclusion Criteria:

* For observational study: health volunteers and cancer patients
* For DC vaccine: patients with solid tumor

Exclusion Criteria:

* leukemia

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Immune status | 5 years

SECONDARY OUTCOMES:
Tumor response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: I-Hsuan A Chen, D.Phil, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan